CLINICAL TRIAL: NCT01584596
Title: Steps Ahead, Adapting Physical Activity Guidelines for the Lower Mississippi Delta Population
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Peter T. Katzmarzyk, Associate Executive Director for Population Science, Professor and Louisiana Public Facilities Authority Endowed Chair, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PBRC 11028
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
Keywords: physical activity; dietary; adults; pedometer; education
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adapted Diet and Physical Activity (Experimental): Adapted diet and physical activity guidelines sessions
  Interventions: Behavioral: Adapted Dietary Guidelines; Behavioral: Adapted Physical Activity Guidelines
- Adapted Diet (Active Comparator): Adapted dietary guidelines sessions
  Interventions: Behavioral: Adapted Dietary Guidelines

INTERVENTIONS:
Behavioral: Adapted Dietary Guidelines — This group will receive dietary counseling to reduce their overall dietary food intake by 100 kcal/day, as prescribed by the dietary guidelines for the prevention of weight gain, and to follow an adapted eating pattern (to be determined from formative research in Phase I research).
  The education sessions will be organized into two phases: an initial adoption phase and a subsequent adherence phase. During the adoption phase, participants will meet for one session per week for the first four weeks. During this session their interim weight will be recorded before they receive their session. During the adherence phase, participants will be contacted by telephone biweekly by a trained interventionist.
Behavioral: Adapted Physical Activity Guidelines — The physical activity education sessions will be organized into two phases: an initial adoption phase and a subsequent adherence phase. The adoption phase will be for 1 hour and 45 minutes for the first 4 weeks with classes occurring once per week in conjunction with the DG education classes. During the adoption phase, participants monitor their own walking using pedometers and attend weekly group meetings to review the previous week's walking behaviors, discuss preferred strategies for success, and set personally relevant and incremental steps/day goals. During the adherence phase (the remaining 8 weeks), participants will continue with their self-monitoring and goal-setting (using their pedometers), with reduced contact with the study interventionists over the telephone (biweekly).
  Other Names: Pedometer
  Arms: Adapted Diet and Physical Activity

SUMMARY:
The Lower Mississippi Delta (LMD) population is characterized by high levels of overweight and obesity, which are the result of long-term disruptions in energy imbalance where dietary energy intake has exceeded energy expenditure associated with physical activity. To address this issue, the overall goal of this project is to determine ways in which the U.S. Department of Health and Human Services and U.S. Department of Agriculture Dietary Guidelines for Americans (2005) physical activity recommendations can be effectively adapted for the LMD population. Phase I of this study was completed in early 2011.

DETAILED DESCRIPTION:
During Phase I, we determined the feasibility of adapting physical activity recommendations by incorporating pedometers (step-counters) as self-monitoring tools within the context of an education program. Lessons learned from the feasibility study have been incorporated into the design of the current proposed Phase II program. This study will be an appropriately powered, randomized controlled effectiveness trial of physical activity and adapted dietary guidelines (DG) eating patterns to reduce unhealthy weight gain. The Steps Ahead study will use the step-based physical activity recommendations identified in Phase I.

Participants will be randomized and orientated into one of two groups. One group will be an adapted DG group who will receive education on the adapted DG guidelines. The second group will be an adapted DG plus physical activity group who will also receive the adapted DG guidelines education plus a physical activity intervention. The diet and physical activity recommendations have been developed to be used as low-intensity interventions in order to ensure maximal sustainability in the population. This intervention will be undertaken in East Baton Rouge parish, an area of the Delta region which contains communities and neighborhoods representative of the broader Delta region.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-64 years
* Body mass index (BMI) 25 to 34.9 kg/m2
* Physically capable of undertaking physical activity
* The capability and willingness to give written informed consent, to understand exclusion criteria, and to accept the randomized group assignment

Exclusion Criteria:

* Blood pressure greater than 159 mmHg systolic or 99 mmHg diastolic
* Total cholesterol greater than or equal to 240 mg/dl with LDL-C greater than or equal to 160 mg/dl or TG levels greater than or equal to 300 mg/dl
* Previously undiagnosed or uncontrolled Type 2 diabetes
* A past history and/or physical examination or laboratory findings of a medical condition including but not limited to chronic or recurrent cardiovascular, respiratory, gastrointestinal, neuromuscular, neurological, or psychiatric conditions.
* Musculoskeletal problems interfering with exercise. Immunodeficiency diseases or a positive HIV test.
* Malignancies in the past 5 years, with the exception of skin cancer therapeutically controlled.
* Any other medical condition or disease that is life-threatening or that can interfere with or be aggravated by exercise
* Pregnant or breastfeeding or plans to become pregnant within the next 4 months.
* Has taken any form of weight loss medication or medications known to affect weight in the past 30 days.
* Have begun taking any new regular prescription medications within the last 3 months (a 3 month stable dose is allowed)
* Planning on starting any new form of medication within the next 4 months
* Being an athlete or highly and regularly physically active (defined as 20 minutes of vigorous activity 3 times per week or 30 minutes of moderate activity 5 times per week)
* Participants not providing adequate accelerometry data i.e. who have not worn the device during waking hours for a full 7 days will be excluded at Visit 3.

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Body weight | Week 0, 1, 2, 3 and 4 and week 12 (termination of intervention)
  Body weight change

SECONDARY OUTCOMES:
Moderate to Vigorous Physical Activity | Week 0 and week 13
  Accelerometer measured moderate to vigocous physical activity levels

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Katzmarzyk, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Harrington DM, Champagne CM, Broyles ST, Johnson WD, Tudor-Locke C, Katzmarzyk PT. Steps ahead: a randomized trial to reduce unhealthy weight gain in the Lower Mississippi Delta. Obesity (Silver Spring). 2014 May;22(5):E21-8. doi: 10.1002/oby.20684. Epub 2014 Jan 25. PMID 24376252
- [Result] Harrington DM, Champagne CM, Broyles ST, Johnson WD, Tudor-Locke C, Katzmarzyk PT. Cardiometabolic risk factor response to a lifestyle intervention: a randomized trial. Metab Syndr Relat Disord. 2015 Apr;13(3):125-31. doi: 10.1089/met.2014.0112. Epub 2015 Jan 8. PMID 25569324
- [Result] Barreira TV, Harrington DM, Schuna JM Jr, Tudor-Locke C, Katzmarzyk PT. Pattern changes in step count accumulation and peak cadence due to a physical activity intervention. J Sci Med Sport. 2016 Mar;19(3):227-231. doi: 10.1016/j.jsams.2015.01.008. Epub 2015 Feb 3. PMID 25687483